CLINICAL TRIAL: NCT03916081
Title: A Phase 2, 4-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-151 Cream 0.05% and ARQ-151 Cream 0.15% Administered QD (Quaque Die) in Adolescent and Adult Subjects With Atopic Dermatitis
Brief Title: Safety and Efficacy of ARQ-151 Cream in Adolescents and Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ-151-212
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Roflumilast Cream 0.05% (Active Comparator): Participants apply roflumilast cream 0.05% QD for 28 days.
  Interventions: Drug: Roflumilast Cream 0.05%
- Roflumilast Cream 0.15% (Active Comparator): Participants apply roflumilast cream 0.15% QD for 28 days.
  Interventions: Drug: Roflumilast Cream 0.15%
- Vehicle Cream (Placebo Comparator): Participants apply vehicle cream QD for 28 days.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Roflumilast Cream 0.05% — Roflumilast 0.05% cream for topical application
  Other Names: ARQ-151
  Arms: Roflumilast Cream 0.05%
Drug: Roflumilast Cream 0.15% — Roflumilast 0.15% cream for topical application
  Other Names: ARQ-151
  Arms: Roflumilast Cream 0.15%
Drug: Vehicle Cream — Inactive vehicle cream matched to roflumilast cream for topical application.
  Arms: Vehicle Cream

SUMMARY:
The study will assess the safety, pharmacokinetics (PK), and efficacy of different doses of roflumilast (ARQ-151) cream (0.05% and 0.15%) vs placebo applied once daily (QD) for 28 days by adolescents and adults with atopic dermatitis.

DETAILED DESCRIPTION:
This is a parallel group, double blind, vehicle-controlled study in which roflumilast cream 0.05% or 0.15% or vehicle is applied QD x 28 days to adolescent and adult subjects with atopic dermatitis. A subset of subjects will have serial PK testing, which will include the first few adolescents and adults enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent or, in the case of adolescents, assent with consent of a parent(s) or legal guardian, as required by local laws.
2. Males and females ages 12 years and older (inclusive) at the time of consent.
3. Clinical diagnosis of active atopic dermatitis for at least 6 months.
4. BSA (Body Surface Area) involvement of at least 2% but no more than 25% at Baseline.
5. vIGA-AD (validated Investigator Global Assessment-Atopic Dermatitis) score of 'mild' ('2') or 'moderate ('3') at Baseline.
6. EASI (Eczema Area and Severity Index) score of ≥ 5 at Baseline.
7. Females of childbearing potential must have a negative serum pregnancy test at Screening and, if sexually active, agree to use birth control throughout the trial.
8. In good health as judged by the Investigator, based on medical history, physical examination, and clinical tests.

Exclusion Criteria:

1. Subjects with any serious medical condition or clinically significant physical examination or test abnormality that would prevent study participation or place the subject at significant risk.
2. Evidence of skin conditions other than AD (atopic dermatitis) that would interfere with evaluation of the effect of the study medication.
3. Pregnant or lactating women or women planning to become pregnant during the study.
4. Known allergies to excipients in ARQ-151 cream.
5. Subjects who cannot discontinue the use of strong P-450 cytochrome inducers or inhibitors .
6. Subjects who are unwilling to refrain from using a tanning bed as well as outdoor tanning or excessive sun exposure.
7. Subjects with unstable AD or who cannot discontinue systemic and/or topical therapies for the treatment of AD.
8. Known or suspected:

   * severe renal insufficiency or moderate to severe hepatic disorders (Child-Pugh B or C)
   * history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or human immunodeficiency virus (HIV))
   * within last 5 years, a history of severe depression, suicidal ideation
9. Previous treatment with ARQ-151.
10. Subjects with a history of chronic alcohol or drug abuse in past 6 months.
11. Current or a history of cancer within 5 years with the exception of fully excised skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
12. Subjects with active infection that requires oral or intravenous administration of antibiotics, antifungal or antiviral agents.
13. Subjects with a history of a major surgery within 8 weeks prior to Baseline or has a major surgery planned during the study.
14. Subjects with any condition which makes them unsuitable for clinical study participation or are family members of the clinical study site, clinical study staff, sponsor, or family members of enrolled subjects.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (20):
- United States (17):
  - Arcutis Clinical Site 25, Scottsdale, Arizona
  - Arcutis Clinical Site 01, San Diego, California
  - Arcutis Clinical Site 19, Hialeah, Florida
  - Arcutis Clinical Site 18, Miami, Florida
  - Arcutis Clinical Site 17, Sanford, Florida
  - Arcutis Clinical Site 16, Boise, Idaho
  - Arcutis Clinical Site 12, Indianapolis, Indiana
  - Arcutis Clinical Site 13, Plainfield, Indiana
  - Arcutis Clinical Site 15, Metairie, Louisiana
  - Arcutis Clinical Site 03, Fridley, Minnesota
  - Arcutis Clinical Site 02, High Point, North Carolina
  - Arcutis Clinical Site 08, Bexley, Ohio
  - Arcutis Clinical Site 23, Pittsburgh, Pennsylvania
  - Arcutis Clinical Site 20, Murfreesboro, Tennessee
  - Arcutis Clinical Site 09, College Station, Texas
  - Arcutis Clinical Site 04, San Antonio, Texas
  - Arcutis Clinical Site 21, Richmond, Virginia
- Canada (3):
  - Arcutis Clinical Site 14, Cobourg, Ontario
  - Arcutis Clinical Site 10, Richmond Hill, Ontario
  - Arcutis Clinical Site 06, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescent (12 to 17 years of age) and adult (≥18 years of age) male and female participants with mild to moderate atopic dermatitis (AD) were enrolled at 3 study sites in Canada and 19 sites in the US.
Period: Overall Study
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Started | 46 | 45 | 45
Completed | 42 | 44 | 42
Not Completed | 4 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1
Not completed — Worsening of AD | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream | Total
Number analyzed (Participants) | 46 | 45 | 45 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (16.98) | 38.0 (16.46) | 42.4 (17.64) | 41.6 (17.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 29 | 93
  Male | 15 | 12 | 16 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 13 | 32
  Not Hispanic or Latino | 36 | 35 | 32 | 103
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 1 | 5 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 14 | 11 | 36
  White | 32 | 24 | 32 | 88
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: score on a scale] — The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
  score on a scale | 8.44 (4.149) | 9.50 (4.097) | 9.20 (3.877) | 9.04 (4.039)
Baseline Body Surface Area (BSA) Score [Mean (Standard Deviation); unit: percentage of body surface area] — The percentage of BSA affected by AD is determined by the subject's hand method, where the subject's hand (including fingers) surface area was assumed to equal 1% of BSA. All AD lesions on a subject were treated including the face, trunk, genitals/skin folds, or limbs (excluding the scalp); the palms and soles were treated but were not counted towards any measurements of BSA.
  percentage of body surface area | 8.4 (7.11) | 9.6 (5.99) | 10.5 (6.62) | 9.5 (6.60)
Baseline Worst Itch Numerical Rating Scale (WI-NRS) Score [Mean (Standard Deviation); unit: score on a scale] — The WI-NRS is a simple, single item scale to assess the participant-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participant experienced in the past 24 hours. Higher scores indicate greater symptom severity.
  score on a scale | 6.48 (1.986) | 6.60 (2.049) | 7.20 (2.106) | 6.76 (2.057)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 4
Description: The least squares (LS) mean (SD) change from baseline in EASI Total Score at Week 4 is reported. The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Time Frame: Baseline and Week 4
Population: All randomized participants with data are included.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 42 | 44 | 44
score on a scale | -6.03 (0.503) | -6.44 (0.492) | -4.84 (0.492)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Change from Baseline in Week 4 EASI Total Score: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.356, MMRM — MMRM = mixed effects model for repeated measures vIGA-AD = validated Investigator Global Assessment scale for Atopic Dermatitis; Change from BL MMRM model includes treatment, visit, vIGA-AD strata, treatment-by-visit interaction as fixed effects and baseline EASI as a covariate; LS Mean Difference vs Vehicle = -1.18, 95% CI 2-sided [-2.983 to 0.619] — Change from BL MMRM model includes treatment, visit, vIGA-AD strata, treatment-by-visit interaction as fixed effects and baseline EASI as a covariate
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Change from Baseline in Week 4 EASI Total Score: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.097, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference vs Vehicle = -1.60, 95% CI 2-sided [-3.382 to 0.178] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage Change From Baseline in EASI Total Score
Description: The LS mean (SD) percentage change from baseline in EASI Total Score at Weeks 1, 2, and 4 is reported. The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: All randomized participants with data are included.
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
percent change
  Week 1: number analyzed (Participants) | 44 | 44 | 44
  Week 1 | -35.77 (4.297) | -34.67 (4.273) | -24.39 (4.279)
  Week 2: number analyzed (Participants) | 42 | 44 | 44
  Week 2 | -54.30 (4.663) | -57.65 (4.567) | -48.48 (4.571)
  Week 4: number analyzed (Participants) | 42 | 44 | 44
  Week 4 | -69.37 (4.643) | -72.32 (4.546) | -55.84 (4.551)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Percent Change from Baseline in Week 1 EASI Total Score: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.248, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -11.37, 95% CI 2-sided [-26.789 to 4.044] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Percent Change from Baseline in Week 1 EASI Total Score: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.349, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -10.28, 95% CI 2-sided [-25.666 to 5.114] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Percent Change from Baseline in Week 2 EASI Total Score: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.912, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -5.82, -22.520% CI 2-sided [-22.520 to 10.880] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Percent Change from Baseline in Week 2 EASI Total Score: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.548, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -9.17, 95% CI 2-sided [-25.686 to 7.341] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Percent Change from Baseline in Week 4 EASI Total Score: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.164, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -13.53, 95% CI 2-sided [-30.157 to 3.097] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Percent Change from Baseline in Week 4 EASI Total Score: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.049, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -16.48, 95% CI 2-sided [-32.921 to -0.048] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change From Baseline in EASI Total Score at Weeks 1 and 2
Description: The LS mean (SD) change from baseline in EASI Total Score at Weeks 1 and 2 is reported. The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Time Frame: Baseline and Weeks 1 and 2
Population: All randomized participants with data are included.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
score on a scale
  Week 1: number analyzed (Participants) | 44 | 44 | 44
  Week 1 | -3.11 (0.416) | -2.77 (0.57) | -2.19 (0.414)
  Week 2: number analyzed (Participants) | 42 | 44 | 44
  Week 2 | -4.80 (0.479) | -5.02 (0.469) | -4.31 (0.470)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Change from Baseline in Week 1 EASI Total Score: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.440, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.92, 95% CI 2-sided [-2.412 to 0.568] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Change from Baseline in Week 1 EASI Total Score: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.875, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.57, 95% CI 2-sided [-2.061 to 0.914] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants Achieving a 50% Decrease From Baseline in EASI Score (EASI-50)
Description: The number of participants with a decrease of at least 50% from the baseline EASI total score is presented. The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease), with positive results indicating an increase from baseline in EASI total score (i.e., increased symptoms) and negative results indicating a decrease from baseline score (i.e., decreased symptoms). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: All randomized participants with ≥1 post-baseline assessment are included (last observation carried forward [LOCF] used for missing data after Week 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
Participants
  Week 1: number analyzed (Participants) | 44 | 44 | 44
  Week 1 | 14 | 11 | 10
  Week 2: number analyzed (Participants) | 44 | 44 | 45
  Week 2 | 27 | 23 | 22
  Week 4: number analyzed (Participants) | 44 | 44 | 45
  Week 4 | 32 | 33 | 25
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-50 at Week 1: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.352, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-50 at Week 1: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.803, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 3: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-50 at Week 2: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.250, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-50 at Week 2: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.756, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 5: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-50 at Week 4: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.097, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-50 at Week 4: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.054, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor

5. Secondary Outcome: Number of Participants Achieving a 75% Decrease From Baseline in EASI Score (EASI-75)
Description: The number of participants with a decrease of at least 75% from the baseline EASI total score is presented. The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease), with positive results indicating an increase from baseline in EASI total score (i.e., increased symptoms) and negative results indicating a decrease from baseline score (i.e., decreased symptoms). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: All randomized participants with ≥1 post-baseline assessment are included (LOCF used for missing data after Week 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
Participants
  Week 1: number analyzed (Participants) | 44 | 44 | 44
  Week 1 | 4 | 6 | 1
  Week 2: number analyzed (Participants) | 44 | 44 | 45
  Week 2 | 8 | 14 | 11
  Week 4: number analyzed (Participants) | 44 | 44 | 45
  Week 4 | 26 | 23 | 14
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-75 at Week 1: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.178, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-75 at Week 1: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.046, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 3: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-75 at Week 2: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.469, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-75 at Week 2: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.446, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 5: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-75 at Week 4: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-75 at Week 4: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.045, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor

6. Secondary Outcome: Number of Participants Achieving a 90% Decrease From Baseline in EASI Score (EASI-90)
Description: The number of participants with a decrease of at least 90% from the baseline EASI total score is presented. The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease), with positive results indicating an increase from baseline in EASI total score (i.e., increased symptoms) and negative results indicating a decrease from baseline score (i.e., decreased symptoms). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI. In some instances, it was not possible to compare roflumilast to vehicle due to low number of cases.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: All randomized participants with ≥1 post-baseline assessment are included (LOCF used for missing data after Week 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
Participants
  Week 1: number analyzed (Participants) | 44 | 44 | 44
  Week 1 | 0 | 1 | 0
  Week 2: number analyzed (Participants) | 44 | 44 | 45
  Week 2 | 1 | 6 | 4
  Week 4: number analyzed (Participants) | 44 | 44 | 45
  Week 4 | 8 | 12 | 8
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-90 at Week 1: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.317, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 2: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-90 at Week 2: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.182, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 3: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-90 at Week 2: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.485, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 4: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-90 at Week 4: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.913, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 5: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-90 at Week 4: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.288, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor

7. Secondary Outcome: Number of Participants Achieving a 100% Decrease From Baseline in EASI Score (EASI-100)
Description: The number of participants with a decrease of 100% from the baseline EASI total score is presented. The EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). The EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease), with positive results indicating an increase from baseline in EASI total score (i.e., increased symptoms) and negative results indicating a decrease from baseline score (i.e., decreased symptoms). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI. In some instances, it was not possible to compare roflumilast to vehicle due to low number of cases.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: All randomized participants with ≥1 post-baseline assessment are included (LOCF used for missing data after Week 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
Participants
  Week 1: number analyzed (Participants) | 44 | 44 | 44
  Week 1 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 44 | 44 | 45
  Week 2 | 1 | 2 | 0
  Week 4: number analyzed (Participants) | 44 | 44 | 45
  Week 4 | 1 | 5 | 1
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-100 at Week 2: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.340, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-100 at Week 2: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.146, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 3: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number Achieving EASI-100 at Week 4: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.967, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number Achieving EASI-100 at Week 4: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.088, Cochran-Mantel-Haenszel; Baseline vIGA-AD was included as stratification factor

8. Secondary Outcome: Mean Change From Baseline in Body Surface Area (BSA) Involvement
Description: The LS mean (SE) change from baseline in BSA involvement at Weeks 1, 2, and 4 is presented. The BSA affected by AD was determined by the subject's hand method, where the subject's hand (including fingers) surface area was assumed to equal 1% of BSA. Negative scores indicate improvement of symptoms, whereas positive scores indicate worsening.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: All randomized participants with data are included.
Measure: Least Squares Mean (Standard Error); unit: percentage of BSA affected
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
percentage of BSA affected
  Week 1: number analyzed (Participants) | 44 | 44 | 44
  Week 1 | -1.19 (0.407) | -1.67 (0.407) | -1.57 (0.405)
  Week 2: number analyzed (Participants) | 42 | 44 | 44
  Week 2 | -2.69 (0.580) | -3.63 (0.570) | -3.29 (0.568)
  Week 4: number analyzed (Participants) | 42 | 44 | 44
  Week 4 | -4.41 (0.658) | -5.10 (0.645) | -4.16 (0.644)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Change from Baseline in BSA Affected at Week 1: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.989, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = 0.38, 95% CI 2-sided [-1.098 to 1.852] — Change from BL MMRM model includes treatment, visit, vIGA-AD strata, treatment-by-visit interaction as fixed effects and baseline BSA as a covariate
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Change from Baseline in BSA Affected at Week 1: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p > 0.999, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.10, 95% CI 2-sided [-1.566 to 1.367] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Change from Baseline in BSA Affected at Week 2: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.966, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = 0.60, 95% CI 2-sided [-1.510 to 2.702] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Change from Baseline in BSA Affected at Week 2: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.999, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.34, 95% CI 2-sided [-2.415 to 1.744] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Change from Baseline in BSA Affected at Week 4: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p > 0.999, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.25, 95% CI 2-sided [-2.624 to 2.119] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Change from Baseline in BSA Affected at Week 4: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.798, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.94, 95% CI 2-sided [-3.285 to 1.398] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Worse Itch Numerical Rating Score (WI-NRS) Score Change
Description: The LS mean (SE) change from baseline in WI-NRS score is presented. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. Higher scores indicate greater symptom severity.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: All randomized participants with data are included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
score on a scale
  Week 1: number analyzed (Participants) | 44 | 44 | 44
  Week 1 | -2.21 (2.13) | -2.46 (0.361) | -1.7 (2.52)
  Week 2: number analyzed (Participants) | 42 | 44 | 44
  Week 2 | -2.46 (0.415) | -2.76 (0.413) | -2.04 (0.408)
  Week 4: number analyzed (Participants) | 42 | 44 | 44
  Week 4 | -3.34 (0.449) | -3.23 (0.444) | -2.73 (0.440)
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Change from Baseline in WI-NRS at Week 1: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.466, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.78, 95% CI 2-sided [-2.075 to 0.506] — Change from BL MMRM model includes treatment, visit, vIGA-AD strata, treatment-by-visit interaction as fixed effects and baseline WI-NRS as a covariate
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Change from Baseline in WI-NRS at Week 1: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.180, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -1.03, 95% CI 2-sided [-2.322 to 0.255] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Change from Baseline in WI-NRS at Week 2: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.967, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.43, 95% CI 2-sided [-1.921 to 1.069] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Change from Baseline in WI-NRS at Week 2: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.684, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.72, 95% CI 2-sided [-2.205 to 0.762] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Change from Baseline in WI-NRS at Week 4: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.856, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.61, 95% CI 2-sided [-2.221 to 1.003] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Change from Baseline in WI-NRS at Week 4: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.932, MMRM; Dunnett's method was used to control for multiple comparisons; LS Mean Difference = -0.51, 95% CI 2-sided [-2.105 to 1.089] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Number of Participants Achieving ≥4-Point Improvement in WI-NRS Pruritus Score
Description: The number of participants achieving a ≥4-point improvement from Baseline in WI-NRS score is presented. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. Higher scores indicate greater symptom severity.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: All randomized participants with data are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 46 | 45 | 45
Participants
  Week 1: number analyzed (Participants) | 41 | 39 | 41
  Week 1 | 11 | 15 | 9
  Week 2: number analyzed (Participants) | 41 | 39 | 42
  Week 2 | 10 | 15 | 16
  Week 4: number analyzed (Participants) | 41 | 39 | 42
  Week 4 | 21 | 17 | 18
Statistical Analysis 1: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number of Participants Achieving a ≥4-Point Improvement from Baseline WI-NRS at Week 1: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.637, Cochran-Mantel-Haenszel; v-IGA-AD included as a stratification factor
Statistical Analysis 2: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.124, Cochran-Mantel-Haenszel; v-IGA-AD included as a stratification factor
Statistical Analysis 3: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number of Participants Achieving a ≥4-Point Improvement from Baseline WI-NRS at Week 2: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.196, Cochran-Mantel-Haenszel; v-IGA-AD included as a stratification factor
Statistical Analysis 4: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p = 0.985, Cochran-Mantel-Haenszel; v-IGA-AD included as a stratification factor
Statistical Analysis 5: Comparison: Roflumilast Cream 0.05% vs Vehicle Cream; Number of Participants Achieving a ≥4-Point Improvement from Baseline WI-NRS at Week 4: Roflumilast Cream 0.05% vs. Vehicle Cream; Test type: Superiority; p = 0.401, Cochran-Mantel-Haenszel; v-IGA-AD included as a stratification factor
Statistical Analysis 6: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; Number of Participants Achieving a ≥4-Point Improvement from Baseline WI-NRS at Week 4: Roflumilast Cream 0.15% vs. Vehicle Cream; Test type: Superiority; p = 0.996, Cochran-Mantel-Haenszel; v-IGA-AD included as a stratification factor

ADVERSE EVENTS:
Time Frame: Up to 32 days
Description: All participants who received ≥1 dose of study intervention are included.
Arm/Group | Roflumilast Cream 0.05% | Roflumilast Cream 0.15% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/46 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Cream 0.05% (N=46) | Roflumilast Cream 0.15% (N=45) | Vehicle Cream (N=45)
Traumatic spinal cord compression (Injury, poisoning and procedural complications) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT03916081/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03916081/SAP_001.pdf